CLINICAL TRIAL: NCT06268275
Title: Comparison of Effects of Scalp Block and Intravenous Esmolol on Hemodynamic Response Following the Skull Pins Application for Elective Supratentorial Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Akkhara Olanvoravuth, Akkhara Olanvoravuth, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HE651314
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hemodynamic Instability
MeSH Terms: interventions — esmolol

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): Receive 30 ml of 0.25% bupivacaine with 1% lidocaine (1:1) with adrenaline 1:200,000 infiltration for 10 minutes before skull pins application.
  Interventions: Procedure: Scalp block
- Group E (Active Comparator): Receive intravenous esmolol 1 mg/kg bolus over 1 minute before skull pins application.
  Interventions: Drug: Esmolol

INTERVENTIONS:
Procedure: Scalp block — Receive 30 ml of 0.25% bupivacaine with 1% lidocaine (1:1) with adrenaline 1:200,000 infiltration for 10 minutes before skull pins application.
  Arms: Group S
Drug: Esmolol — Receive Intravenous esmolol 1 mg/kg bolus over 1 minute before skull pins application
  Arms: Group E

SUMMARY:
The goal of this clinical trial is to compare hemodynamic response (MAP, SBP, DBP and HR) between scalp block and intravenous esmolol while skull pins application in patients undergoing elective supratentorial craniotomy under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* BMI 18-30 kg/m2
* American Society of Anesthesiologists (ASA) status I-III
* Elective supratentorial craniotomy under general anesthesia
* Required application of skull pins

Exclusion Criteria:

* Poor controlled hypertensive condition (Baseline BP ≥ 160/110 mmHg)
* Thrombocytopenia / Coagulopathy
* Preoperative atrioventricular block (More than 2nd degree AV block)
* Emergency surgery
* Posterior fossa / Intracranial aneurysm surgery
* Pregnancy
* Chronic use of pain control
* Contraindication to beta-blockers
* Allergy to the drugs used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
MAP | Baseline, 1 minute before skull pins, then 30 sec, 60 sec, 90 sec, 120 sec, 180 sec and 300 sec after skull pins
  Mean arterial pressure
SBP | Baseline, 1 minute before skull pins, then 30 sec, 60 sec, 90 sec, 120 sec, 180 sec and 300 sec after skull pins
  Systolic blood pressure
DBP | Baseline, 1 minute before skull pins, then 30 sec, 60 sec, 90 sec, 120 sec, 180 sec and 300 sec after skull pins
  Diastolic blood pressure
HR | Baseline, 1 minute before skull pins, then 30 sec, 60 sec, 90 sec, 120 sec, 180 sec and 300 sec after skull pins
  Heart rate

SECONDARY OUTCOMES:
BIS | Baseline, 1 minute before skull pins, then 30 sec, 60 sec, 90 sec, 120 sec, 180 sec and 300 sec after skull pins
  Bispectral index
Cumulative postoperative opioids consumption | 6 hours and 24 hours postoperatively
  Opioids consumption
Postoperative adverse events | Within first 24 hours postoperatively
  Incidence (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Khon Kaen University, Khon Kaen, Naimuang, Muang, Thailand

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: Researchers who required more information for further study

REFERENCES:
- [Background] Fukuda S, Warner DS. Cerebral protection. Br J Anaesth. 2007 Jul;99(1):10-7. doi: 10.1093/bja/aem140. PMID 17573393
- [Background] Li J, Gelb AW, Flexman AM, Ji F, Meng L. Definition, evaluation, and management of brain relaxation during craniotomy. Br J Anaesth. 2016 Jun;116(6):759-69. doi: 10.1093/bja/aew096. Epub 2016 Apr 27. PMID 27121854
- [Background] Colley PS. Blunting the hemodynamic response to skull-pin placement. Anesth Analg. 1997 Apr;84(4):942. doi: 10.1097/00000539-199704000-00056. No abstract available. PMID 9085997
- [Background] Singh G, Arimanikam G, Lionel KR, Smita V, Yadav B, Arulvelan A, et al. Comparison of Dexmedetomidine Infusion versus Scalp Block with 0.5% Ropivacaine to Attenuate Hemodynamic Response to Skull Pin Insertion in Craniotomy: A Prospective, Randomized Controlled Trial. J Neuroanaesth Crit Care. 2021 Sep;08(03):180-6.
- [Background] Bharne S, Bidkar PU, Badhe AS, Parida S, Ramesh AS. Comparison of intravenous labetalol and bupivacaine scalp block on the hemodynamic and entropy changes following skull pin application: A randomized, open label clinical trial. Asian J Neurosurg. 2016 Jan-Mar;11(1):60-5. doi: 10.4103/1793-5482.165801. PMID 26889282
- [Background] Yang SH, Liu R. Cerebral Autoregulation. In: Primer on Cerebrovascular Diseases [Internet]. Elsevier; 2017 [cited 2022 Jun 10]. p. 57-60.
- [Background] Jellish WS, Theard MA, Cheng MA, Leonetti JP, Crowder CM, Tempelhoff R. The effects of clonidine premedication and scalp infiltration of lidocaine on hemodynamic responses to laryngoscopy and skull pin head-holder insertion during skull base procedures. Skull Base. 2001 Aug;11(3):169-76. doi: 10.1055/s-2001-16605. PMID 17167618
- [Background] Misra S, Koshy T, Unnikrishnan KP, Suneel PR, Chatterjee N. Gabapentin premedication decreases the hemodynamic response to skull pin insertion in patients undergoing craniotomy. J Neurosurg Anesthesiol. 2011 Apr;23(2):110-7. doi: 10.1097/ANA.0b013e3181da3c3b. PMID 20479668
- [Background] Koo CH, Jeon S, Kim J, Ryu JH. The effects of intravenous dexmedetomidine on hemodynamic response in patients undergoing skull-pin head-holder application during neurosurgery - A meta-analysis of randomized controlled trials. Clin Neurol Neurosurg. 2020 Aug;195:105939. doi: 10.1016/j.clineuro.2020.105939. Epub 2020 May 20. PMID 32480196
- [Background] Doblar DD, Lim YC, Baykan N, Frenette L. A comparison of alfentanil, esmolol, lidocaine, and thiopental sodium on the hemodynamic response to insertion of headrest skull pins. J Clin Anesth. 1996 Feb;8(1):31-5. doi: 10.1016/0952-8180(95)00169-7. PMID 8695076
- [Background] Agarwal A, Sinha PK, Pandey CM, Gaur A, Pandey CK, Kaushik S. Effect of a subanesthetic dose of intravenous ketamine and/or local anesthetic infiltration on hemodynamic responses to skull-pin placement: a prospective, placebo-controlled, randomized, double-blind study. J Neurosurg Anesthesiol. 2001 Jul;13(3):189-94. doi: 10.1097/00008506-200107000-00002. PMID 11426091
- [Background] Geze S, Yilmaz AA, Tuzuner F. The effect of scalp block and local infiltration on the haemodynamic and stress response to skull-pin placement for craniotomy. Eur J Anaesthesiol. 2009 Apr;26(4):298-303. doi: 10.1097/EJA.0b013e32831aedb2. PMID 19262392
- [Background] Altaf I, Banday J, Naaz S, Ozair E, Punetha P, Challam K. A randomized control trial on comparative effect of scalp nerve block using levobupivacaine versus fentanyl on the attenuation of pain and hemodynamic response to pin fixation. Bali J Anesthesiol. 2021;5(2):66.
- [Background] Yang X, Ma J, Li K, Chen L, Dong R, Lu Y, Zhang Z, Peng M. A comparison of effects of scalp nerve block and local anesthetic infiltration on inflammatory response, hemodynamic response, and postoperative pain in patients undergoing craniotomy for cerebral aneurysms: a randomized controlled trial. BMC Anesthesiol. 2019 Jun 1;19(1):91. doi: 10.1186/s12871-019-0760-4. PMID 31153358
- [Background] Hagan KB, Bhavsar S, Raza SM, Arnold B, Arunkumar R, Dang A, Gottumukkala V, Popat K, Pratt G, Rahlfs T, Cata JP. Enhanced recovery after surgery for oncological craniotomies. J Clin Neurosci. 2016 Feb;24:10-6. doi: 10.1016/j.jocn.2015.08.013. Epub 2015 Oct 21. PMID 26474504
- [Background] Watts R, Thiruvenkatarajan V, Calvert M, Newcombe G, van Wijk RM. The effect of perioperative esmolol on early postoperative pain: A systematic review and meta-analysis. J Anaesthesiol Clin Pharmacol. 2017 Jan-Mar;33(1):28-39. doi: 10.4103/0970-9185.202182. PMID 28413270
- [Background] Gelineau AM, King MR, Ladha KS, Burns SM, Houle T, Anderson TA. Intraoperative Esmolol as an Adjunct for Perioperative Opioid and Postoperative Pain Reduction: A Systematic Review, Meta-analysis, and Meta-regression. Anesth Analg. 2018 Mar;126(3):1035-1049. doi: 10.1213/ANE.0000000000002469. PMID 29028742
- [Background] Morais VBD, Sakata RK, Huang APS, Ferraro LHDC. Randomized, double-blind, placebo-controlled study of the analgesic effect of intraoperative esmolol for laparoscopic gastroplasty. Acta Cir Bras. 2020 Jun 5;35(4):e202000408. doi: 10.1590/s0102-865020200040000008. eCollection 2020. PMID 32555939
- [Background] Kang JK, Yoo SH, Chung JH, Kim NS, Jung HS, Seo YH, Chun HR, Gong HY, Son HD, Kim AJ. Dosing study of esmolol for reducing hemodynamic changes during lightwand intubation. Anesth Pain Med (Seoul). 2020 Oct 30;15(4):417-423. doi: 10.17085/apm.19067. PMID 33329844
- [Background] Sola C, Dadure C, Choquet O, Capdevila X. Nerve Blocks of The Face. NYSORA [Internet]. 2018 Sep 17 [cited 2022 Jun 10]; Available from: https://www.nysora.com/techniques/head-and-neck-blocks/nerve-blocks-face/
- [Background] Hockey B, Leslie K, Williams D. Dexamethasone for intracranial neurosurgery and anaesthesia. J Clin Neurosci. 2009 Nov;16(11):1389-93. doi: 10.1016/j.jocn.2009.03.007. Epub 2009 Aug 7. PMID 19665383
- [Background] Uribe AA, Stoicea N, Echeverria-Villalobos M, Todeschini AB, Esparza Gutierrez A, Folea AR, Bergese SD. Postoperative Nausea and Vomiting After Craniotomy: An Evidence-based Review of General Considerations, Risk Factors, and Management. J Neurosurg Anesthesiol. 2021 Jul 1;33(3):212-220. doi: 10.1097/ANA.0000000000000667. PMID 31834247